CLINICAL TRIAL: NCT02947594
Title: Half-life of Plasma Phytosterols in Very Low Birth Weight Preterm Infants With Parenteral Nutrition-associated Cholestasis
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Virgilio Paolo Carnielli, MD, Phd, Professor of Neonatal Pediatrics at Polytechnical University of Marche (Ancona, Italy), Università Politecnica delle Marche
Other Study IDs: DG469
Record Dates: First submitted 2016-09-06; First posted 2016-10-28 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Parenteral nutrition-associated cholestasis (PNAC) is one of the most common complications resulting from administration of parenteral nutrition in neonates. Excess intravenous intake of vegetable oil-based lipid emulsions containing phytosterols is felt to be a major contributing factor. To date, no information is available on plasma phytosterols half-lives in very-low-birth-weight (VLBW) preterm infants with PNAC. In a prospective cohort study, plasma phytosterols (campesterol, stigmasterol and sitosterol) of VLBW preterm infants with PNAC will be measured by gas chromatography-mass spectrometry (GC-MS) during PN administration and also after the stop of intravenous lipid infusion. Plasma phytosterols half-lives will be calculated from the monoexponential decay curves. Blood samples will be weekly collected from 1st to 12th week of life during routine metabolic tolerance analysis or gas-analysis in order to avoid burden of additional phlebotomy. Samples will be collected in ethylenediaminetetraacetic acid-tubes and immediately centrifugated. Plasma will be stored in pyrogallol added-tubes at -20°C until analysis. Saponification reaction will be done using 5-alpha-cholestane as internal standard.

ELIGIBILITY:
Inclusion Criteria:

* 24 weeks < gestational age < 32 weeks;
* 500 g ≤ birth weight < 1250 g;
* parenteral nutrition with vegetable oil-based lipid emulsions from the first hours of life;
* diagnosis of cholestasis during vegetable oil-lipid infusion (plasma conjugated bilirubin value > 1 mg/dl)
* parental consent;

Exclusion Criteria:

* severe malformations;
* inborn errors of metabolism;
* severe congenital sepsis;
* normal liver functions (plasma conjugated bilirubin under 1 mg/dl during vegetable oil-lipid infusion).

Ages: 24 Weeks to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (24 < gestational age < 32 weeks; 500 g ≤ birth weight < 1250 g) with parenteral nutrition-associated cholestasis.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change of plasma phytosterol concentrations in preterm infants during parenteral nutrition and after only intravenous lipid stopping | 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77 and 84 days
  Plasma campesterol, stigmasterol and sitosterol concentrations will be measured at 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77 and 84 days from PN started. Plasma phytosterol concentrations will be measured by gas chromatography-mass spectrometry. Calibration curves will be used to calculate the phytosterol plasma concentrations (mg/L).

SECONDARY OUTCOMES:
Liver dysfunction in preterm infants will be defined by conjugated bilirubin values from blood samples over 1 mg/dl | Routinely checked at 7 and 42 days of life. Additional measure of conjugated bilirubin will be performed after 15 days if the value continues to be higher than 1 mg/dl.
  Eligibility of preterm infants will be related to liver function. Conjugated bilirubin value from blood sample is a good sign of hepatic function. The threshold value was defined to 1 mg/dl. Just preterm infants who will have conjugated bilirubin values more of 1 mg/dl will be included in the study. Conjugated bilirubin will be measured at 7 and 42 days of life on routine care. When the conjugated bilirubin value will be higher than 1 mg/dl, the analysis will be repeated every 15 days until it returns under the threshold value (1 mg/dl). Parenteral nutrition-associated cholestasis will be only diagnosed in patients with pathological values of conjugated bilirubin (over 1 mg/dl) during vegetable oil-lipid infusion.
Plasma phytosterols half-lives | We will able to measure the plasma phytosterol half-lives (days) after the analysis of 3 or more blood samples collected from the stop of lipid infusion to 84 days of life
  Plasma phytosterol half-lives (days) will be measured using 3 or more plasma phytosterol concentrations calculated after only lipid stopping. Half-life of plasma phytosterols will be calculated from monoexponential decay curves.

REFERENCES:
- [Background] Zaloga GP. Phytosterols, Lipid Administration, and Liver Disease During Parenteral Nutrition. JPEN J Parenter Enteral Nutr. 2015 Sep;39(1 Suppl):39S-60S. doi: 10.1177/0148607115595978. Epub 2015 Jul 15. PMID 26177665
- [Background] Savini S, D'Ascenzo R, Biagetti C, Serpentini G, Pompilio A, Bartoli A, Cogo PE, Carnielli VP. The effect of 5 intravenous lipid emulsions on plasma phytosterols in preterm infants receiving parenteral nutrition: a randomized clinical trial. Am J Clin Nutr. 2013 Aug;98(2):312-8. doi: 10.3945/ajcn.112.056556. Epub 2013 Jun 12. PMID 23761482
- [Background] Nghiem-Rao TH, Tunc I, Mavis AM, Cao Y, Polzin EM, Firary MF, Wang X, Simpson PM, Patel SB. Kinetics of phytosterol metabolism in neonates receiving parenteral nutrition. Pediatr Res. 2015 Aug;78(2):181-9. doi: 10.1038/pr.2015.78. Epub 2015 Apr 21. PMID 25897540
- [Background] El Kasmi KC, Anderson AL, Devereaux MW, Vue PM, Zhang W, Setchell KD, Karpen SJ, Sokol RJ. Phytosterols promote liver injury and Kupffer cell activation in parenteral nutrition-associated liver disease. Sci Transl Med. 2013 Oct 9;5(206):206ra137. doi: 10.1126/scitranslmed.3006898. PMID 24107776
- [Background] Weingartner O, Teupser D, Patel SB. The Atherogenicity of Plant Sterols: The Evidence from Genetics to Clinical Trials. J AOAC Int. 2015 May-Jun;98(3):742-749. doi: 10.5740/jaoacint.SGEWeingartner. Epub 2015 May 19. PMID 25942705
- [Background] Bhattacharyya AK, Connor WE, Lin DS, McMurry MM, Shulman RS. Sluggish sitosterol turnover and hepatic failure to excrete sitosterol into bile cause expansion of body pool of sitosterol in patients with sitosterolemia and xanthomatosis. Arterioscler Thromb. 1991 Sep-Oct;11(5):1287-94. doi: 10.1161/01.atv.11.5.1287. PMID 1911714
- [Background] Lin HJ, Wang C, Salen G, Lam KC, Chan TK. Sitosterol and cholesterol metabolism in a patient with coexisting phytosterolemia and cholestanolemia. Metabolism. 1983 Feb;32(2):126-33. doi: 10.1016/0026-0495(83)90216-0. PMID 6827984
- [Background] Salen G, Tint GS, Shefer S, Shore V, Nguyen L. Increased sitosterol absorption is offset by rapid elimination to prevent accumulation in heterozygotes with sitosterolemia. Arterioscler Thromb. 1992 May;12(5):563-8. doi: 10.1161/01.atv.12.5.563. PMID 1576118
- [Background] Ellegard L, Sunesson A, Bosaeus I. High serum phytosterol levels in short bowel patients on parenteral nutrition support. Clin Nutr. 2005 Jun;24(3):415-20. doi: 10.1016/j.clnu.2005.01.001. PMID 15896428